CLINICAL TRIAL: NCT03679156
Title: Retinal Pigment Epithelial Characteristics in Eyes With Neovascular Age-related Macular Degeneration Following Long-term Treatment With Anti Neovascular Endothelial Growth Factor
Status: Completed | Type: Observational
Sponsor: Hospital Hietzing (Other)
Responsible Party: Principal Investigator, Dr. Clara Wernigg, Dr., Hospital Hietzing
Other Study IDs: RPE characteristics
Record Dates: First submitted 2018-09-19; First posted 2018-09-20 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: Neovascular Age-related Macular Degeneration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: OCT — Patients were recruited, visual acuity and optical coherence tomography Pictures were taken

SUMMARY:
Purpose:

To assess retinal pigment epithelial (RPE) and retinal structural changes in eyes with neovascular age-related macular degeneration (AMD) treated with anti-vascular endothelial growth factor (anti-VEGF) during long-term follow-up and to evaluate morphological markers potentially influencing prognosis.

Methods:

18 patients (18 eyes) with neovascular AMD were recruited subsequent to completion the Avastin Versus Lucentis in Age Related Macular Degeneration (MANTA) study following a mean period of 84 months (range: 69-93 months). After receiving a loading dose of 3 intravitreal anti-VEGF injections subsequent to baseline of the MANTA study, patients were treated as-needed [pro re nata (PRN)]. Functional and morphological changes were assessed using spectral domain optical coherence tomography (SD-OCT).

ELIGIBILITY:
Inclusion Criteria:

* Inclusion and exclusion criteria corresponded to the criteria of the MANTA study

Exclusion Criteria:

* Inclusion and exclusion criteria corresponded to the criteria of the MANTA study

Ages: 66 Years to 98 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Initially 55 Participants were included in the Avastin Versus Lucentis in Age Related Macular Degeneration (MANTA) trial [16]. These patients received a loading dose of 3 intravitreal injections of anti-VEGF and were subsequently treated as-needed [pro re nata (PRN)] [16]. From that study population we recruited for another long term follow up visit. Of these patients 9 (16%) were excluded due to missed visits, another 14 patients (25%) died before the last study visit and 14 former participants (25%) did not approve further study participation.
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2016-05-30 (Actual); Primary Completion 2016-11-02 (Actual); Study Completion 2017-04-15 (Actual)

PRIMARY OUTCOMES:
visual acuity | 93 months
  visual acuity testing was performed

IPD SHARING:
Plan to Share IPD: No